CLINICAL TRIAL: NCT02652286
Title: Pulmonary Artery Harmonic Ace+7 Energy Sealing in VATS Lobectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 15.270
Record Dates: First submitted 2015-12-07; First posted 2016-01-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Lung Cancer
Keywords: VATS; Energy sealing
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Harmonic Ace+7 (Other): Pulmonary artery sealing with Harmonic Ace+7 in VATS lobectomy
  Interventions: Device: HARMONIC ACE+7

INTERVENTIONS:
Device: HARMONIC ACE+7 — Pulmonary artery sealing with Harmonic Ace+7 in VATS lobectomy in humans

SUMMARY:
Video-assisted thoracic surgery (VATS) anatomical lung resection provides an effective minimally invasive treatment strategy for stage I and II lung cancer. VATS lobectomy is associated with significantly less postoperative atrial fibrillation, blood transfusion, renal failure, and other complications when compared with lobectomy via thoracotomy.

Although VATS lobectomy has been proven to be effective and safe in experienced hands, it is not devoid of risk. Intra-operative surgical complications can be at times catastrophic. Complications include: pulmonary vascular injuries (Pulmonary artery (PA), pulmonary vein) necessitating urgent conversion to open thoracotomy and even death. Causes of conversion included PA injury, difficult anatomy, bulky/calcified lymph nodes, and technical problems including stapler misfire. PA injury alone constituted 37.5% of all conversions. Proper dissection of all tissue around PA branches is sometime difficult especially in the presence of adhesions or large, calcified lymph nodes and may increase the risk of vascular injury.

Currently, in spite of being a safe and effective technique in experienced hands, a minority of anatomical pulmonary resections are being performed by VATS. In an analysis utilizing the Nationwide Inpatient Sample (NIS) database in the United States, only 15% of anatomical lung resections were performed by VATS.

The technical difficulty and danger of VATS lobectomy is directly related to PA branch manipulation, stapling and division. PA manipulation is the main hesitation of many thoracic surgeons regarding the adoption of VATS lobectomy. We believe that if we can decrease the manipulation and dissection required by the surgeon on the PA branches, we can make these procedures safe and therefore more prevalent for anatomical pulmonary resections.

DETAILED DESCRIPTION:
This study consists of evaluating the safety and efficacy of energy sealing lobar PA branches for lobectomy in humans. All patients planned to undergo a lobectomy by VATS at the CHUM - Hôpital Notre-Dame will be approached. In our institution, lobectomies are either done open (thoracotomy) or by minimally invasive approach, known as VATS (video assisted thoracoscopic surgery). This decision is based on the surgeon, tumor size, tumor localization and patient characteristics. Only patients already planned for a VATS lobectomy will be approached. Potential patients will be selected by going over the operation request forms. Patients booked for a VATS lobectomy will be approached either in the preoperative clinic or the day before surgery, when admitted. Aim is to recruit 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned to undergo a VATS lobectomy at the CHUM-Hopital Notre-Dame

Exclusion Criteria:

* Age > 18 years old
* Inability to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
All patients will be assessed for effective intra-operative pulmonary arterial branch vessel sealing. It will be measured visually by the presence or lack of vessel sealing failure | 30 days
  All cases will be videotaped with a thoracosocpic 10 mm, 30 degree camera placed through the chest tube insertion site in order to evaluate the problems in cases of seal failure. All patients will have 4-0 prolene with SH needle ready for use on the sterile field in case there is a sealing failure that needs to be fixed.
  Additionally, all patients are routinely crossmatched for 2 units of packed red blood cells (as per standard pre-operative orders).

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre Hospitalier de l'Université
Locations (1):
- CHUM-Notre Dame Hospital, Montreal, Quebec, Canada